CLINICAL TRIAL: NCT04938557
Title: Automated Insulin Delivery Amongst Pregnant Women With Type 1 Diabetes
Acronym: AiDAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other); University of Cambridge (Other); University of Leeds (Other); University of Edinburgh (Other); University of Glasgow (Other); King's College London (Other); Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 240380
Record Dates: First submitted 2021-05-18; First posted 2021-06-24 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Diabetes
Keywords: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: An open-label, multi-centre, randomized, two-arm parallel group trial
Masking Description: This is an unblinded trial. Both participants and their clinical care team will be aware of the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An Automated Closed-loop Insulin Delivery (AiD) System. (Experimental): The intervention being evaluated in this trial is automated closed-loop insulin delivery (AiD). The closed-loop system comprises of three components: an insulin pump, a continuous glucose monitor (CGM) and a computer-based model predictive control (MPC) algorithm to compute information from the CGM into a recommended insulin dose.
  Interventions: Device: Automated closed-loop insulin delivery (AiD)
- A Standard Insulin Delivery System (Active Comparator): This can include either: an insulin pump (Continuous Subcutaneous Insulin Infusion - CSII) or multiple daily injections (MDI) without closed-loop.
  Interventions: Device: A standard insulin delivery system

INTERVENTIONS:
Device: Automated closed-loop insulin delivery (AiD) — Closed-loop systems are designed to deliver insulin in response to CGM glucose levels and may help to improve glucose control above and beyond what is currently achievable using insulin pumps, injections and CGM without AiD.
  Arms: An Automated Closed-loop Insulin Delivery (AiD) System.
Device: A standard insulin delivery system — Self-directed insulin delivery for pregnant women with T1D, which is insulin pump or MDI.
  Arms: A Standard Insulin Delivery System

SUMMARY:
Evaluation of the biomedical and psychosocial impact of automated Closed-Loop (Artificial Pancreas) insulin delivery in women with type 1 diabetes during pregnancy

DETAILED DESCRIPTION:
An open-label, multi-centre, randomized, two-arm parallel group trial comparing automated closed-loop and standard insulin delivery.

124 pregnant women between 18 and 45 years of age with Type 1 Diabetes of at least 12 months' duration on standard insulin delivery (CSII or MDI) will be recruited through outpatient antenatal diabetes clinics. Women fulfilling the eligibility criteria will be randomized to automated insulin delivery (AiD) or to continue standard patient-directed insulin delivery (CSII or MDI) without AiD. The study will take place within the home and NHS antenatal clinical settings.

Additional blood samples for the research will be obtained at the 24th and 34th week of pregnancy and questionnaires will also be completed by the participant at the 34th week of pregnancy. Following this we will collect information on the birth.

25 of the woman randomised to the closed loop insulin delivery system will also be interviewed to gain more information on, among other things, their existing diabetes management practices, everyday work and family lives and their experience with the device.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 45 years of age (inclusive).
2. A diagnosis of type 1 diabetes (T1D), as defined by WHO for at least 12 months.
3. A viable pregnancy confirmed by ultrasound, up to 13 weeks and 6 days gestation.
4. Currently on intensive insulin therapy (≥3 injections or CSII).
5. Willingness to use the study devices throughout the trial.
6. HbA1c level ≥48 mmol/mol (≥6.5%) at booking (first antenatal contact) and ≤86 mmol/mol (≤10%) at point of randomization.
7. Able to provide informed consent.
8. Have access to email.

Exclusion Criteria:

1. Non-type 1 diabetes.
2. Any other physical or psychological disease which, in the opinion of the investigator, is likely to interfere with the normal conduct and interpretation of the study results e.g. untreated coeliac disease or untreated hypothyroidism.
3. Current treatment with drugs known to interfere with glucose metabolism as judged by the investigator such as high dose systemic corticosteroids, non-selective beta-blockers and MAO inhibitors.
4. Known or suspected allergy against insulin.
5. Women with advanced nephropathy (eGFR <45), severe autonomic neuropathy, uncontrolled gastroparesis or severe proliferative retinopathy, as judged by the investigator, that is likely to interfere with the normal conduct of the study and interpretation of study results.
6. Very good or very poor glycaemic control i.e. first antenatal HbA1c <48 mmol/mol (<6.5%) and current HbA1c >10% (>86 mmol/mol). Women who enter pregnancy with HbA1c >10% (>86 mmol/mol) may participate if they achieve HbA1c ≤10% (≤86 mmol/mol) before randomization.
7. Total daily insulin dose 1.5 IU/kg.
8. Severe visual or hearing impairment.
9. Unable to speak and understand English.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The time spent with glucose levels between 3.5-7.8 mmol/L based on CGM measures (Time In Range TIR 3.5-7.8mmol/L) | Between 16 weeks gestation and delivery - an average of 18 weeks
  The primary outcome is the percentage of time spent with glucose levels between 3.9-7.8 mmol/L based on CGM levels between 16 weeks gestation and delivery.as compared with standard self-directed insulin delivery in pregnant women with T1D.

SECONDARY OUTCOMES:
CGM glucose measures | Between 16 weeks gestation and delivery - an average of 18 weeks
  The time spent with CGM glucose levels above and below target range, using the mean CGM glucose and CGM glucose variability measures (CV, SD).
CGM glucose index (Low) | Between 16 weeks gestation and delivery - an average of 18 weeks
  The Low Blood Glucose Index (LBGI)
CGM glucose index (High) | Between 16 weeks gestation and delivery - an average of 18 weeks
  High Blood Glucose Index (HBGI) measures
HbA1c testing (Maternal) | Blood samples will be collected at baseline, 24-26 weeks, 34-36 weeks
  To assess the change of HbA1c in the maternal level.
Diabetic ketoacidosis. | An average of 24 weeks
  The frequency and severity of diabetic ketoacidosis
Severe hypoglycaemia episodes. | An average of 24 weeks
  The frequency and severity of hypoglycaemia episodes defined as CGM glucose levels <3.5 mmol/L (level 1 hypoglycaemia) and <2.8 mmol/L (level 2 hypoglycaemia) for at least 15 minutes. Distinct episodes must be separated for at least 30 minutes.
The number and severity of episodes of adverse device effect. | <24 weeks gestation until delivery - an average of 16 weeks
  Adverse events including pregnancy loss, stillbirth, neonatal death
Hospital length of stay (maternal). | Between 13 and 40 weeks - an average of 24 weeks
  Hospital length of stay (all admissions including the delivery admission)
Mode of delivery | At >34 weeks (delivery)
  How the infant is delivered, for example: vaginal, instrumental, elective caesarean section and emergency caesarean section)
Gestational age at delivery | At >34 weeks (delivery)
  The gestational age at delivery and indication for any preterm delivery (<37 weeks). Measured in years.
Infant birth weight (LGA) | At >34 weeks (delivery)
  Infant birth weight (customised birth weight percentile, incidence of large for gestational age (LGA).
Infant birth weight (SGA). | At >34 weeks (delivery)
  Infant birth weight (customised birth weight percentile, incidence of small for gestational age (SGA).
Neonatal morbidity (hypoglycaemia, jaundice, respiratory distress). | Between delivery and 40 weeks - an average of 6 weeks
  Neonatal morbidity including treatment for neonatal hypoglycaemia, neonatal jaundice and respiratory distress.
Neonatal intensive care unit (NICU) admission. | NICU admission after 24 hours
  Neonatal intensive care unit (NICU) admission >24 hours
Hospital length of stay (infant). | Between delivery and 40 weeks - an average of 6 weeks
  Hospital length of stay for the infant

CONTACTS AND LOCATIONS:
Overall Officials: Helen Murphy, Principal Investigator — University of East Anglia
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Lawton J, Kimbell B, Closs M, Hartnell S, Lee TTM, Dover AR, Reynolds RM, Collett C, Barnard-Kelly K, Hovorka R, Rankin D, Murphy HR. Listening to Women: Experiences of Using Closed-Loop in Type 1 Diabetes Pregnancy. Diabetes Technol Ther. 2023 Dec;25(12):845-855. doi: 10.1089/dia.2023.0323. Epub 2023 Nov 7. PMID 37795883
- [Derived] Rankin D, Hart RI, Kimbell B, Barnard-Kelly K, Brackenridge A, Byrne C, Collett C, Dover AR, Hartnell S, Hunt KF, Lee TTM, Lindsay RS, McCance DR, McKelvey A, Rayman G, Reynolds RM, Scott EM, White SL, Hovorka R, Murphy HR, Lawton J. Rollout of Closed-Loop Technology to Pregnant Women with Type 1 Diabetes: Healthcare Professionals' Views About Potential Challenges and Solutions. Diabetes Technol Ther. 2023 Apr;25(4):260-269. doi: 10.1089/dia.2022.0479. Epub 2023 Feb 27. PMID 36662589